CLINICAL TRIAL: NCT03097458
Title: Enhancing Adjustment to Parental Cancer: Short-term Counselling for Families. A Randomized, Wait-list Controlled Intervention Study
Brief Title: Enhancing Adjustment to Parental Cancer: Short-term Counselling for Families
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: propatient Forschungsstiftung (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PP-16-07
Record Dates: First submitted 2017-03-10; First posted 2017-03-31 (Actual); Last update posted 2020-07-07 (Actual); Status verified 2020-07

CONDITIONS: Psychological Adjustment; Cancer
Keywords: Counselling for Families; Parental cancer; Psychological distress and adjustment
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Intervention Model Description: Randomized wait-list control design (cross-over).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Counselling (Experimental): short-term counselling for families
  Interventions: Behavioral: Short-term Counselling for Families
- Wait-list control group (No Intervention): Wait-list control group

INTERVENTIONS:
Behavioral: Short-term Counselling for Families — Counselling for Families which can take up to 6 weeks, with regular meetings under the guidance of a trained psychotherapist.
  Arms: Counselling

SUMMARY:
A parental cancer diagnosis challenges the family's stability and the parent-child relationship. It may impact the children's well-being, so that about one third of them develop clinically relevant levels of psychological distress. Psycho-oncological family-based counselling programs have been shown to elevate children's and parents' well-being. However, there is still a dearth of familial health services in Switzerland, which has also been recognized by the Swiss National Cancer Program (2011-2017).

This study aims to implement and evaluate a short-term family counselling intervention at the Cancer Center of the University Hospital Basel. The primary objective of the study is the enhancement of adjustment to the parental cancer diagnosis. The study seeks secondary to determine the feasibility of the short-term counselling Intervention.

DETAILED DESCRIPTION:
This study ist designed as a randomized controlled wait-list Intervention study, which aims to implement and evaluate a short-term family counselling intervention at the Cancer Center of the University Hospital Basel. The study will be divided into two stages: Stage 1 serves as the preparatory work phase, where the intervention manual will be developed as well as the implementation strategy into the hospital. In stage 2 the intervention will be evaluated, with an interim analysis to test for feasibility. The primary objective of the study is the enhancement of adjustment (family, parents and children) to the parental cancer diagnosis. The study seeks secondary to determine the feasibility of the short-term counselling intervention in the Swiss medical setting and to identify predictors for families with continuing psychosocial adjustment problems.

ELIGIBILITY:
Inclusion Criteria:

* Informed Consent as documented by signature
* Diagnosis of any kind of cancer, inclusive relapse, within the last year with an expected survival of at least 8 months
* Married, cohabiting or single parent
* At least one child between 1-5 - 18 years
* German speaking

Exclusion Criteria:

* The diagnosis is more than 1 year ago
* Diagnosed patients (parent) not living with their children
* Diagnosed patients without custody of their children

Min Age: 18 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2017-02-04 (Actual); Primary Completion 2019-09-01 (Actual); Study Completion 2019-09-01 (Actual)

PRIMARY OUTCOMES:
Change of children's quality of life on the health-related quality of life questionnaire (KINDL) | 6 weeks (change between baseline and week 6)
  Enhancement of children's quality of life from T1 (baseline) to T2 (6 weeks) compared to the wait-list control group.
Change of children's behavioral-emotional functioning on the Strengths and Difficulties Questionnaire (SDQ) | 6 weeks (change between baseline and week 6)
  Enhancement of children's behavioral-emotional functioning from T1 (baseline) to T2 (6 weeks) compared to the wait-list control group.
Change of parent's mental health on the Hospital Anxiety and Depression Scale (HADS) | 6 weeks (change between baseline and week 6)
  Enhancement of parent's mental health from T1 (baseline) to T2 (6 weeks) compared to the wait-list control group.
Change of family functioning on the Family Adaptability and Cohesion Evaluation Scale (FACES IV) | 6 weeks (change between baseline and week 6)
  Enhancement of family functioning from T1 (baseline) to T2 (6 weeks) compared to the wait-list control group.
Change of relationship quality on the relationship questionnaire (Partnerschaftsfragebogen PFB) | 6 weeks (change between baseline and week 6)
  Enhancement of relationship quality from T1 (baseline) to T2 (6 weeks) compared to the wait-list control group.

SECONDARY OUTCOMES:
Number of participants willing to participate in the counselling | Through study completion, an average of 2 years
  Secondary outcome will be to determine whether a short-term counselling intervention is feasible in the Swiss medical setting by collecting the number of participants willing to participate.
Sociodemographic characteristics (i.e. age, gender, education) of the participants willing to participate in the counselling with the sociodemographic questionnaire | Through study completion, an average of 2 years
  Collecting sociodemographic characteristics of the population willing to participate with the sociodemographic questionnaire
Medical history characteristics (i.e. cancer diagnosis, cancer treatment) of the participants willing to participate in the counselling with the medical history questionnaire | Through study completion, an average of 2 years
  Collecting medical history of the population willing to participate with the medical history questionnaire
Dropout rate during the recruitment and intervention procedure | Through study completion, an average of 2 years
  Secondary outcome will be to determine whether a short-term counselling intervention is feasible in the Swiss medical setting by collecting dropout rate during the recruitment and intervention procedure.
Client satisfaction on the Client Satisfaction Questionnaire (CSQ-8) | Measures assessed after 6 weeks
  German Version of the Client Satisfaction Questionnaire: Fragebogen zur Messung der Patientenzufriedenheit (ZUF-8) will be used to measure client's intervention satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Corinne Urech, Dr. phil., Principal Investigator — University Hospital, Basel, Switzerland
Locations (1):
- University Hospital Basel, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: No